CLINICAL TRIAL: NCT00880334
Title: Randomized Study of Docetaxel +/- Vandetanib in Metastatic TCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Toni Choueiri, MD, Assistant Professor of Medicine, Harvard Medical School, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-116; NCT00378794 (obsolete NCT alias)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Transitional Cell Carcinoma; Bladder Cancer
Keywords: TCC; Zactima; docetaxel; ZD6474; taxotere
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Docetaxel; vandetanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vandetanib & Docetaxel (Experimental): vandetanib orally and Docetaxel intravenously
  Interventions: Drug: Docetaxel; Drug: vandetanib
- Placebo and Docetaxel (Active Comparator): Placebo orally and docetaxel intravenously
  Interventions: Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: Docetaxel — Given intravenously on Day 1 of each 21-day cycle
  Other Names: Taxotere
Drug: vandetanib — taken orally once a day, every day
  Other Names: ZD6474; Zactima
  Arms: vandetanib & Docetaxel
Drug: Placebo — Taken orally once a day every day
  Arms: Placebo and Docetaxel

SUMMARY:
In this research study the investigators are looking to see if the combination of docetaxel plus Vandetanib is effective in the treatment of metastatic transitional cell carcinoma (TCC). Docetaxel is a chemotherapy drug that kills cancer cells that are dividing. It is widely used in TCC. Vandetanib is a drug that is believed to stop new blood vessels from forming around cancer cells. The combination of docetaxel and Vandetanib has been studied in people with lung cancer and found to be helpful in killing cancer cells. Thus, this study is looking at people with TCC, to see if the combination of docetaxel plus Vandetanib is better or worse then docetaxel alone.

DETAILED DESCRIPTION:
* Because no one knows which of the study options is best, and all of the options are considered equally likely to work, participants will be randomized into one of two study groups: docetaxel plus Vandetanib or docetaxel plus placebo.
* Each treatment cycle lasts three weeks during which time the participant will be taking Vandetanib or placebo once a day, every day. On Day 1 of each cycle (a cycle is 21 days), participants will receive docetaxel as an infusion through a vein in the arm over one hour.
* On Day 1 of every cycle the following tests and procedures will be performed: physical exam and blood tests. On day 1 and on Day 8 of the first cycle only, participants will have an ECG. Every 6-9 weeks (every 2 to 3 cycles), the participants tumor will be assessed by x-ray, CT scan, bone scan, and/or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed TCC. Mixed histologies are allowed as long as the predominant histology is TCC.
* Must have received chemotherapy treatment for TCC and have stage IV TCC at the time of study entry. 1-3 prior systemic chemotherapeutic or investigational treatment regimens for TCC are allowed. Patient with more regimens than the ones allowed may be included at the discretion of the Overall Principal Investigator if it is felt that the regimen has shown minimal activity and toxicity and will not influence prior or subsequent therapies. Specifically, participants must meet one or more of the following criteria: a) Progression after treatment with a regimen that includes a platinum salt (e.g. carboplatin or cisplatin) for Stage IV disease OR b) Disease recurrence within two years (from the date of last dose of chemotherapy or surgery until day the informed consent is signed) after neoadjuvant or adjuvant treatment with a regimen that includes a platinum salt.
* Measurable or evaluable disease, as defined by RECIST. If all sites of measurable or evaluable disease have been irradiated, one site must have demonstrated growth after irradiation.
* Adequate contraceptive method for subjects with reproductive potential (females with reproductive potential must have a negative serum pregnancy test within 7 days of study entry).
* ECOG PS 0 or 1
* 18 years of age or older

Exclusion Criteria:

* History of treatment of TCC (in any setting-neoadjuvant, adjuvant or for metastatic disease) with docetaxel. Patients treated with prior paclitaxel (Taxol) are eligible.
* History of treatment with a VEGF-axis active agent, including antibodies to VEGF, antibodies to VEGF receptors, or VEGF receptor tyrosine kinase inhibitors.
* Laboratory results as outlined in the protocol
* Evidence of uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
* Clinically significant cardiac event such as myocardial infarction; NHYA classification of heart disease >2 within three months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia
* History of arrhythmia, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation which is symptomatic or requires treatment (CTCAE Grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication.
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age.
* Presence of left bundle branch block (LBBB)
* QTc with Bazett's correction that is unmeasurable, or 480 msec or greater on screening ECG. If a subject has a QTc of 480msec or greater on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the subject to be eligible for the study.
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function.
* Hypertension not controlled by medical therapy
* Currently active diarrhea
* Women who are currently pregnant or breast feeding
* Receipt of any investigational agent, chemotherapy or radiation therapy within 21 days prior to Study Day 1
* Any unresolved non-hematologic toxicity greater than CTCAE grade 1 from previous anti-cancer therapy (other than alopecia).
* Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.
* Grade 2 or greater peripheral neuropathy
* Previous or current malignancies within the last 3 years, with the exception of in situ carcinoma of the cervix, adequately treated carcinoma of the skin, small renal masses, and adequately treated localized prostate cancer. Other cancers that are highly likely to be cured (cure rate of 75% or greater) may be included at the discretion of the Overall Principal Investigator.
* History of severe hypersensitivity reaction to drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2006-09; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choueiri TK, Ross RW, Jacobus S, Vaishampayan U, Yu EY, Quinn DI, Hahn NM, Hutson TE, Sonpavde G, Morrissey SC, Buckle GC, Kim WY, Petrylak DP, Ryan CW, Eisenberger MA, Mortazavi A, Bubley GJ, Taplin ME, Rosenberg JE, Kantoff PW. Double-blind, randomized trial of docetaxel plus vandetanib versus docetaxel plus placebo in platinum-pretreated metastatic urothelial cancer. J Clin Oncol. 2012 Feb 10;30(5):507-12. doi: 10.1200/JCO.2011.37.7002. Epub 2011 Dec 19. PMID 22184381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from February 2007 through May 2010.
Pre-assignment Details: There were 7 cancelled patients who were randomized but did not receive treatment.
Groups:
- Vandetanib and Docetaxel: Docetaxel: Given intravenously on Day 1 of each 21-day cycle Vandetanib: taken orally once a day, every day
- Placebo and Docetaxel: Docetaxel: Given intravenously on Day 1 of each 21-day cycle Placebo: Taken orally once a day every day
  Eligible participants were allowed to crossover to single agent vandetanib.
Period: Randomized Phase
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Started | 74 | 75
Eligible & Treated | 70 | 72
Completed | 70 | 35
Not Completed | 4 | 40
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Inadequate Labs | 1 | 1
Not completed — Brain Metastasis | 0 | 1
Not completed — Crossover Participants | 0 | 37
Period: Crossover Phase
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Started | 0 | 37 (Only participants randomized to placebo and docetaxel potentially received crossover treatment.)
Completed | 0 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all eligible and treated patients.
Groups:
- Vandetanib & Docetaxel: Docetaxel: Given intravenously on Day 1 of each 21-day cycle Vandetanib: taken orally once a day, every day
- Placebo and Docetaxel: Docetaxel: Given intravenously on Day 1 of each 21-day cycle Placebo: Taken orally once a day every day
- Total: Total of all reporting groups
Arm/Group | Vandetanib & Docetaxel | Placebo and Docetaxel | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 39 | 71
  >=65 years | 38 | 33 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 48 | 49 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 61 | 67 | 128
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the time between randomization and documented disease progression (PD) per RECIST 1.0 criteria or death, or is censored at time of last disease assessment. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Disease evaluations occurred at week 6 and 12 and thereafter every 3 cycles/9 weeks on treatment and every 3 months in follow-up. Participants were followed until PD, death or lost to follow-up. Median survival follow-up was 12 months (range 1-26).
Population: The analysis dataset is comprised of all eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 70 | 72
months | 2.56 [1.81 to 3.06] | 1.58 [1.48 to 3.09]
Statistical Analysis 1: Comparison: Vandetanib and Docetaxel vs Placebo and Docetaxel; The study was designed with 80% power to detect 60% improvement in median PFS from 18 to 28.8 weeks (Vandetanib+docetaxel/Placebo+docetaxel hazard ratio of 0.625) with the addition of Vandetanib while maintaining an overall significance level of 5% in a one-sided test. This assumed exponential distribution of events, accrual of 1.75 patients per week (7-8 patients per month) for 78 weeks with 34 weeks of additional follow-up (112 weeks total). Full information was 118 PFS events; Test type: Superiority or Other; p = 0.939, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.69 to 1.49]

2. Secondary Outcome: Grade 3-5 Toxicity Rate
Description: Grade 3-5 toxicity rate is the percentage of participants experiencing maximum grade of all toxicity types of grade 3-5 with any attribution on treatment during the randomized phase.
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Median treatment duration for this study cohort approximated 2 cycles (range 1-31).
Population: The analysis dataset is comprised of all eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 70 | 72
percentage of participants | 73 [61 to 83] | 57 [45 to 69]

3. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined from date of randomization to date of death or censored at the date the patient was last known alive.
Time Frame: Off treatment, patients were followed for survival information every 6 months (±1 month) until death,up to 2 years after discontinuing therapy, or until lost to follow-up. Median survival follow-up for the study cohort was 12 months (95% CI: 9-18 months).
Population: The analysis dataset is comprised of all eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 70 | 72
months | 5.85 [5.22 to 7.00] | 7.03 [5.19 to 10.41]
Statistical Analysis 1: Comparison: Vandetanib and Docetaxel vs Placebo and Docetaxel; Test type: Superiority or Other; p = .873, Log Rank; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.81 to 1.79]

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as the percentage of participants who achieved a confirmed overall partial response (PR) or complete response (CR) using RECIST criteria on treatment during the randomized phase. Patients without measurable disease only at baseline are included, based on status of non-target lesions.Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease evaluations occurred at week 6 and 12 and thereafter every 3 cycles/9 weeks on treatment. Median treatment duration for this study cohort approximated 2 cycles (range 1-31).
Population: The analysis dataset is comprised of all eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 70 | 72
percentage of participants | 7.1 [2.4 to 15.9] | 11.1 [4.9 to 20.8]
Statistical Analysis 1: Comparison: Vandetanib and Docetaxel vs Placebo and Docetaxel; Test type: Superiority or Other; p = 0.56, Fisher Exact

5. Post Hoc Outcome: Disease Control Rate
Description: Disease control rate is defined as the percentage of participants with confirmed overall Stable Disease (SD) or better using RECIST 1.0 criteria which parallels absence of disease progression (PD) on treatment during the randomized phase. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Patients without measurable disease only at baseline are included, based on status of non-target lesions.
Time Frame: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 70 | 72
percentage of participants | 51 [39 to 64] | 42 [30 to 54]
Statistical Analysis 1: Comparison: Vandetanib and Docetaxel vs Placebo and Docetaxel; Test type: Superiority or Other; p = 0.31, Fisher Exact

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment on the randomized and crossover phases from time of first dose and up to day 30 post-treatment. Median treatment duration for the randomized study cohort was 2 cycles (range 1-31 cycles). Median treatment duration for the crossover study cohort was 2 cycles (range 1-23 cycles).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with vandetanib treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with vandetanib treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3. No further data is available to specify classification of other beyond the general term.
Groups:
- Placebo and Docetaxel-Crossover: Docetaxel: Given intravenously on Day 1 of each 21-day cycle Vandetanib: taken orally once a day, every day
Arm/Group | Vandetanib and Docetaxel | Placebo and Docetaxel | Placebo and Docetaxel-Crossover
Serious Adverse Events (participants affected / at risk) | 42/70 | 26/72 | 6/37
Other Adverse Events (participants affected / at risk) | 22/70 | 12/72 | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib and Docetaxel (N=70) | Placebo and Docetaxel (N=72) | Placebo and Docetaxel-Crossover (N=37)
Allergic reaction (Immune system disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Creatinine (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 6 | 4 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
GI-other (Gastrointestinal disorders) | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 3 | 0
Infection Gr0-2 neut, bladder (Infections and infestations) | 0 | 1 | 0
Infection Gr 0-2 neut, blood (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 1 | 1 | 0
Infection w/ gr 3-4 neut, blood (Infections and infestations) | 0 | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 0 | 0
Infection w/ unk ANC bladder (Infections and infestations) | 1 | 0 | 0
Infection w/ unk ANC peritoneal cavity (Infections and infestations) | 0 | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Leukocytes (Investigations) | 5 | 7 | 0
Lymphopenia (Investigations) | 4 | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 2 | 0 | 0
Neutrophils (Investigations) | 10 | 10 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
PTT (Investigations) | 1 | 0 | 0
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
QTc interval (Investigations) | 1 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin-other (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 0 | 0 | 1
Nausea (General disorders) | 0 | 0 | 1
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib and Docetaxel (N=70) | Placebo and Docetaxel (N=72) | Placebo and Docetaxel-Crossover (N=37)
Abdomen, pain (Gastrointestinal disorders) | 1 | 0 | 0
Alkaline phosphatase (Investigations) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bilirubin (Investigations) | 1 | 0 | 1
Bronchopulmonary, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Constitutional, other (General disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 6 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dry eye syndrome (Eye disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Edema head and neck (General disorders) | 1 | 0 | 0
Edema limb (General disorders) | 3 | 1 | 0
Edema trunk/genital (General disorders) | 2 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Fatigue (General disorders) | 9 | 6 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Fever w/o neutropenia (General disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
GI-other (Gastrointestinal disorders) | 1 | 0 | 0
Head/headache (Nervous system disorders) | 1 | 0 | 0
Hematologic-other (Blood and lymphatic system disorders) | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 1 | 0 | 0
Infection w/ gr3-4 neut, bladder (Infections and infestations) | 0 | 1 | 0
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Leukocytes (Investigations) | 1 | 1 | 0
Lymphopenia (Investigations) | 1 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 1 | 0
Muco/stomatitis by exam, stomach (Gastrointestinal disorders) | 1 | 0 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 0
Neurologic-other (Nervous system disorders) | 1 | 0 | 0
Neuropathy-motor (Nervous system disorders) | 1 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 2 | 2 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pelvic, pain (Reproductive system and breast disorders) | 1 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Respiratory tract hemorrhage NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rigors/chills (General disorders) | 2 | 0 | 0
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Taste disturbance (Nervous system disorders) | 3 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Urinary hemorrhage NOS (Renal and urinary disorders) | 2 | 0 | 0
Vision-blurred (Eye disorders) | 1 | 0 | 0
AST, SGOT (Investigations) | 0 | 0 | 1
ALT, SGPT (Investigations) | 0 | 0 | 1
Alkaline phosphatase (Investigations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hemorrhage-other (Vascular disorders) | 0 | 0 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes